CLINICAL TRIAL: NCT07275424
Title: Open-Label, Single-Arm Phase 2a Pilot Study to Evaluate the Safety and Tolerability of a Daily Subcutaneous Dose of Elamipretide in Older Adults
Brief Title: Study of Healthy Aging and Physical Function With Elamipretide
Acronym: SHAPE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: David Marcinek (Other)
Collaborators: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor-Investigator, David Marcinek, Professor, University of Washington
Organization: University of Washington (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00023162
Record Dates: First submitted 2025-10-15; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Aging, Healthy
Keywords: healthspan; healthy aging; mobility; cognitive function
MeSH Terms: interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide; Benzyl Alcohol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Safety and tolerability of daily subcutaneous injection of elamipretide (Other): single arm ELAM intervention
  Interventions: Drug: Elamipretide will be supplied as a sterile 5.0 mL single-patient, multi-dose glass vial containing 3.75 mL of elamipretide solution (elamipretide [80 mg/mL], phosphate buffer, and benzyl alcohol)

INTERVENTIONS:
Drug: Elamipretide will be supplied as a sterile 5.0 mL single-patient, multi-dose glass vial containing 3.75 mL of elamipretide solution (elamipretide [80 mg/mL], phosphate buffer, and benzyl alcohol) — Primary Study Objective To evaluate the safety and tolerability of daily subcutaneous injections of elamipetide for 4 weeks in adults aged 65-80
  Secondary Objective To assess inflammatory biomarker changes with 4-week daily injection of elamipetide on healthy aging To assess the skeletal muscle health in older subjects with lower aerobic capacity (cardiovascular health) To assess cognitive function changes with 4-week SC daily injection of elamipetide

SUMMARY:
This study will utilize a daily dose of elamipetide for 4 weeks and will screen a sufficient number of subjects for 30 subjects to enroll in the study. The planned duration of the study includes baseline measurement, followed by 4 weeks intervention period, a midpoint (2week ±3days) check-in phone interview, and post intervention visits that mirror the baseline visits. After the last injection, subjects will enter the 2-week follow-up period, concluded by the end-of-study contact.

DETAILED DESCRIPTION:
This study will be a Phase 2a, open-label, single-arm study enrolling older adults subjects with lower function. The primary objective of this study is to evaluate the safety and tolerability of elamipretide, given as daily subcutaneous injection over 4 weeks. Secondary endpoints will test whether the administration of elamipretide results in changes in blood biomarkers of inflammation and improved cognitive and mobility functional performance in an older adult population. This study will be conducted in strict compliance with the protocol, current Good Clinical Practice (GCP) and all Food and Drug Administration (FDA) guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥65 and ≤80 years
2. VO2peak ≤ 37.3ml/kg/min for men and ≤ 25.7ml/kg/min for women as evidence of lower mitochondrial function
3. Are ambulatory and able to perform activities of daily living without assistance
4. Have sufficient venous access for clinical blood draw
5. Willing and able to self-administer injections or have a willing caregiver who is able to administer injections.
6. Speak and read English
7. Have no established daily exercise routine and are not participating in any exercise training program or physical hobby (i.e. dance, martial arts, yoga) and agree to not start any such activities during the course of study participation
8. Willing to avoid the following medications during the course of the study:

Anti-seizure medications

* Coenzyme Q10, creatine, L-carnitine, and other supplements intended to increase muscle mass, energy or function
* Muscle relaxants
* Systemic steroid or immunosuppressive use
* Opioids (regular use of > 10 mg/day morphine equivalents) 9. No known allergies/adverse effects from Fexofenadine 10. Provide documentation of informed consent

Exclusion Criteria:

1. Have significant disease(s) or condition(s) which, in the opinion of the investigator, may put the subject at risk because of their participation in the study or may influence either the results of the study or the subject's ability to participate in the study
2. Presence of severe renal disease (eGFR <30 mL/min) or hepatic disease (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] >2x the upper limit of normal) as evidenced by laboratory results at Screening.
3. Have a history of rhabdomyolysis
4. Have been hospitalized within 3 months prior to screening for major atherosclerotic events (e.g., myocardial infarction, target-vessel revascularization, coronary bypass surgery or stroke) or other major medical condition (as deemed by the primary investigator)
5. Are currently enrolled in a clinical study involving an investigational product or non- approved use of a drug or device or concurrently enrolled in any other type of medical research judged to be scientifically or medically incompatible with this study
6. Have participated within the last 30 days of screening visit in a clinical study involving an investigational product.

   -

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of daily subcutaneous injections of elamipetide: Number of participants with treatment-related adverse events and Number of participants completed 4 weeks of injection | 4 week

SECONDARY OUTCOMES:
blood inflammation markers | up to 5 months from first enrollment
  levels of BDNF, VEGF, IGF-1, IL-6
blood inflammation marker | up to 5 months from first enrollment
  level of TNF-a
Delta 6 minute walk test | 4-6 weeks after enrollment
  Change in distance walked in 6 minutes following 4 weeks of intervention
Delta cognitive function score | 4-6 weeks after enrollment
  MoCA to access cognitive function from different domains. MoCA scale is 0-30 with scores >26 indicating normal cognitive function. This is measured by a scale the higher means better function. Trail marking A&B time faster is better; Stroop timed test for attention, processing speed, and executive control.
Delta skeletal muscle strength | 4-6 weeks from enrollment
  The investigators will measure the change in muscle strength on a 1 rep knee extensor assay following 4 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: David Marcinek, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be published and listed on clinical trial.gov